CLINICAL TRIAL: NCT01235650
Title: Prevalence of Inadvertent Hyperventilation During Intraoperative Anesthetic Care
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Joseph D. Tobias, Chairman Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Other Study IDs: IRB10-00390
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Spinal Fusion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spinal fusion: Patients who underwent complex surgical procedures (spinal fusions) which necessitated arterial line placement and intermittent arterial blood gas analysis

SUMMARY:
This is a retrospective chart review of patients undergoing spinal fusion surgery to see the prevalence of hyperventilation.

DETAILED DESCRIPTION:
Retrospective review of the operative schedules to identify patients who have undergone spinal fusion with placement of an arterial cannula for intermittent arterial blood gas analysis. The intraoperative records will be retrospectively reviewed. The following demographic data will be recorded: age, weight, gender, and co-morbid medical conditions. Ventilatory parameters at the time of ABG analysis will include (respiratory rate and tidal volume). ABG data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent complex surgical procedures (spinal fusions) which necessitated arterial line placement and intermittent arterial blood gas analysis

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Spinal fusion patients
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Incidence of inadvertent hyperventilation | Day 1